CLINICAL TRIAL: NCT04303351
Title: The Relationship Between Periodontitis and Atherosclerotic-related Arterial Stenosis in the Chinese Population
Brief Title: Periodontitis and Atherosclerotic-related Arterial Stenosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ZF2019-010
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Atherosclerosis of Artery
Keywords: arterial stenosis; periodontitis; atherosclerosis; risk factors
MeSH Terms: conditions — Periodontitis; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — All the blood samples will be stored in the biological resource centre of the our research centre after written informed consent obtained from all subjects who voluntarily participated in this clinical study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 0-9 missing teeth: participants with 0-9 missing teeth
- 10-19 missing teeth: participants with 10-19 missing teeth
- 23-31 missing teeth: participants with 23-31 missing teeth
- Edentulous: participants with no teeth

SUMMARY:
This study aimed to evaluate the association between periodontitis and atherosclerosis of the cerebral vasculature in the Chinese population.

DETAILED DESCRIPTION:
Periodontitis has been demonstrated as a risk factor for ischaemic stroke in several clinical studies. Atherosclerosis of the cerebral vasculatureis an important pathological process causing ischaemic stroke. The investigator's study aims to investigate the relationship between tooth loss(used as a surrogate of periodontal disease) and atherosclerotic-related arterial stenosis in the Chinese population. An estimated 1,000 participants that underwent cerebral angiography at Guangdong Provincial Hospital of Chinese Medicine between Apirl 2020 and January 2022 will be recruited in this trial. Arterial stenosis features of each participants will be collected based on the results of digital subtraction angiography (DSA). The missing teeth counts of each participant will be collected and some of them will recieved comprehensive periodontal examination. Besides, blood samples will be collected in order to investigate the serum inflammatory markers(CRP,WBC,albumin,IL-6,IL-10). The relationship between tooth loss and atherosclerotic-related arterial stenosis will be analysed by regression models adjusted for conventional risk factors (sex,age, obesity,smoking,Alcohol drinking,diabetes,hypertension,hyperuricaemia,hyperhomocysteinaemia)

ELIGIBILITY:
Inclusion Criteria:

1. subjects who underwent cerebral angiography at Guangdong Provincial Hospital of Chinese Medicine from April 2020 to December 2021
2. subjects who voluntarily participated in this study and provided informed consent.

Exclusion Criteria:

1. intracranial and extracranial artery stenosis caused by vascular inflammation, systemic connective tissue disease, and muscle fibre structure hypoplasia
2. inability to cooperate with the investigation
3. intracranial aneurysm and cerebral arteriovenous malformation confirmed by cerebral angiography
4. receipt of periodontal treatment in the previous 24 months.

Ages: 18 Years to 98 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population are people who underwent cerebral angiography at Guangdong Provincial Hospital of Chinese Medicine from April 2020 to April 2022 and meat the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
The relationship between atherosclerotic-related stenosis in different brain arteries and tooth loss categories | 1 day
  The arteries of the brains will be partitioned into the following segments: common carotid artery (CCA), internal carotid arteries (ICA, C1-C7), the external carotid artery (ECA), the anterior cerebral artery (ACA, A1-A2), the middle cerebral artery (MCA, M1-M2), the posterior cerebral artery (PCA), the basilar artery (BA), the vertebral artery (VA,V1-V4) and the subclavicular artery (SUB) .The chi-square test and Fisher's exact test will be used, as appropriate, to estimate the relationship between tooth loss and stenosis distributed in different branches

SECONDARY OUTCOMES:
The relationship between the severity of artery stenosis and tooth loss categories | 1 day
  The degree of vascular stenosis will be categorized into five group: no stenosis, mild stenosis, moderate stenosis, severe stenosis and occlusion. Ordinal logistic regression will be performed to analyse the relationship between the tooth loss categories and the degrees of artery stenosis.